CLINICAL TRIAL: NCT05905822
Title: DIetary plAnt Extracts, Colonic MicrObes, and Apoe geNetics Interactions stuDy
Acronym: DIAMOND
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Collaborators: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Other Study IDs: 319832
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease Risks; Microbiome; APOE genotype; Metabolism; Cognition
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary sample Stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospectively genotyped participants: These participants will be advertised to in the local area. They will be genotyped for their APOE genotype, and then the stool sample will be collected.
- Database participants: Participants from the previously genotyped cohort "Early sleep and circadian markers of Alzheimer's disease: the impact of APOE-ε4 on circadian rhythm and sleep-wake homeostasis in humans" (Reference: 2017/18-135) who have consented to be contacted will be contacted to collect a stool sample.

SUMMARY:
This study will involve donating a salivary sample and a faecal (stool) sample. These will be analysed in the laboratory to determine the forms of the APOE gene you are carrying (your APOE genotype) and the response of the bacteria in your colon to reactive compounds extracted from edible plants (dietary bioactives).

DETAILED DESCRIPTION:
In an ageing population, the incidence of dementia is rapidly increasing and poses a significant financial, societal, and above all, personal burden. Aside from ageing, the type of APOE gene an individual carries (their APOE genotype) is the greatest risk factor for the development of cognitive decline. It has been shown that the APOE genotype of an individual influences the types of bacteria present in the colon. The bacteria which reside in the colon have recently emerged as a significant contributor to nutrition and health and have been suggested to influence brain functioning through complex connections between the gut and the brain.

Nutrition is considered important for brain function throughout life, and findings from recent laboratory and human observational studies have suggested that reactive compounds extracted from edible plants (dietary bioactives) can not only improve brain function, but they can change the function and composition of gut bacteria. Dietary bioactives are a range of natural compounds found in great concentrations within fruits and vegetables which influence the body. An example of a dietary bioactive is a group of compounds known as polyphenols. These polyphenols are described as antioxidants and are found in various foods, including berries, tea, and cocoa.

There have been no previous studies looking at the impact of dietary bioactives on the microbiome of each APOE genotype and the metabolites produced by each of these bacteria. We aim with the current study to identify how dietary bioactives from a range of plant tissue could influence gut bacteria present and the metabolites produced by the bacteria in each APOE group, and the compounds produced by these bacteria.

What will the study involve? Once we have established a potentially suitable participant, they will be sent a salivary sampling kit. Depending on the genotype, age and sex, participants will be requested to donate a stool sample. The stool will be processed in a colon model with cocoa polyphenol added.

The study involves the following stages:

1. Online screening, consenting, and collection of basic information
2. Collection of a salivary sample in person at the Clinical Research Facility or home and return to the labs via pre-paid postal mail.
3. Confirmation of eligibility to donate stool samples.
4. Collection of stool samples on the same day as sample collection. Returning the sample in person or through the pre-paid postal system.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years old or aged 55+ years old
* Fluent in written and spoken English and capacity to consent
* Availability to take part in the study

Exclusion Criteria:

* Participants will be excluded from donating if they have been diagnosed with any gastrointestinal conditions such as inflammatory bowel disease.
* They will also be excluded if they have a diagnosis of any form of dementia or severe cognitive impairment.
* They currently consume a high flavonoid intake defined as >15 portions of flavonoid rich food per day.
* History or MRI evidence of brain damage, including significant trauma, stroke, learning difficulties or serious neurological disorder, including a loss of consciousness for more than 24 hours.
* Currently smoking or ceased smoking less than 6 months ago.
* Chronic fatigue syndrome, liver disease, diabetes mellitus, or gall bladder abnormalities.
* History of alcohol or drug dependency.
* Clinically diagnosed psychiatric disorder.
* Currently a participant or have been a participant in any other study involving an investigational product within the last 4 weeks.
* Received a COVID-19 diagnosis within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults who fit the above inclusion and exclusion criteria. Able to donate a stool and salivary sample.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Whether there is a significant difference between the in vitro metabolism of flavan-3-ols using a human colon model | 09/2025
  Participants will be genotyped for their APOE genotype. They will then be requested to donate a stool sample. This stool sample will be run through a colon.model inoculated with flavan-3-ols to determine whether there is a significant difference between the genotypes. Flavan-3-ol metabolism will be measured with LCMS
Determine whether there are significant differences between the composition of the gut microbiome of each APOE genotype. | 09/2025
  Participants will be genotyped for their APOE genotype. Their stool sample will then have its gut microbiome analysed. Metagenomic techniques will be utilised to analyse the microbiome

CONTACTS AND LOCATIONS:
Overall Officials: David Vauzour, PhD, Principal Investigator — University of East Anglia
Locations (1):
- Norwich and Norfolk University Hospital Clinical Research Facility, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raulin AC, Doss SV, Trottier ZA, Ikezu TC, Bu G, Liu CC. ApoE in Alzheimer's disease: pathophysiology and therapeutic strategies. Mol Neurodegener. 2022 Nov 8;17(1):72. doi: 10.1186/s13024-022-00574-4. PMID 36348357
- [Result] Seals RR Jr, Morrow RM, Kuebker WA. The dentist's role in Texas high school mouthguard programs. Tex Dent J. 1984 Oct;101(10):6-9. No abstract available. PMID 6593891